CLINICAL TRIAL: NCT04579614
Title: Performance Feedback in Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: London School of Economics and Political Science (Other)
Responsible Party: Principal Investigator, Felipe Lobelo, Physician Program Director, Epidemiology, Public Health, and Preparedness, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1535959-1
Record Dates: First submitted 2020-09-09; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: Flu Vaccination Provision; Performance Feedback; Variable Goal Setting; Flu Vaccination Success Rate; Health Care Providers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Providers are randomized to receive one of three designs of performance feedback, related to their rate of successful flu vaccinations among total flu opportunities
Who Masked: Participant
Masking Description: Providers do not know that that multiple arms of performance feedback designs exist for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Organizational Target (Active Comparator): Providers are shown the flu success performance rate of their team (a "pod," or group of providers who practice together), in comparison to their own, and with the organizational target. These updates and targets are sent bi-weekly.
  Interventions: Behavioral: The Impact of Performance Feedback and Variable Goal Setting on Flu Vaccination Success Rates of Providers
- Achievable Target (Experimental): Providers are shown the flu success performance rate of their team (a "pod," or group of providers who practice together), in comparison to their own. They will receive a static and achievable target based on their previous year's flu vaccination success rate.
  Interventions: Behavioral: The Impact of Performance Feedback and Variable Goal Setting on Flu Vaccination Success Rates of Providers
- Variable (Experimental): Providers are shown the flu success performance rate of their team (a "pod," or group of providers who practice together), in comparison to their own. They will receive a variable target that will fluctuate bi-weekly, based on their previous bi-weekly flu vaccination success rate.
  Interventions: Behavioral: The Impact of Performance Feedback and Variable Goal Setting on Flu Vaccination Success Rates of Providers

INTERVENTIONS:
Behavioral: The Impact of Performance Feedback and Variable Goal Setting on Flu Vaccination Success Rates of Providers — A given provider will be involved in the study for a maximum of 6 months. This will involve, at the most frequent, the delivery of weekly performance feedback.
  The performance feedback will be delivered using standard approaches already in place in the organization and there will not be a period of seeking out participants for enrollment.
  Providers will receive performance feedback bi-weekly for the duration of the study period.

SUMMARY:
The Southeast Permanente Medical Group (TSPMG) at Kaiser Permanente Georgia provides performance feedback to its providers. The performance feedback designs can vary and change over time in terms of targets, summary statistics, included measures, and frequency of delivery. The TSPMG health services research group seek to compare different performance feedback designs to identify which are most effective at contributing to performance improvement.

The research team will randomly assign providers into different performance feedback conditions, as specified in the protocol. Providers will receive performance feedback through the standard mechanism in which it is conveyed by their supervisor.

The objective is to investigate how to design performance feedback for providers to best motivate and support them in improving performance along with existing strategic priorities for care delivery.

The reserach team will test alternative designs of performance feedback that vary on the following dimension:

1) targets for comparison of one's own performance

DETAILED DESCRIPTION:
The Southeast Permanente Medical Group (TSPMG) provides performance feedback to its providers. The performance feedback designs can vary and change over time in terms of targets, summary statistics, included measures, and frequency of delivery. The TSPMG health services research team will seek to compare different performance feedback designs to identify which are most effective at contributing to performance improvement. .

The research team will randomly assign providers into different performance feedback conditions, as specified in the protocol. Providers will receive performance feedback through the standard mechanism in which it is conveyed by their supervisor.

The objective is to investigate how to design performance feedback for providers to best motivate and support them in improving performance along with existing strategic priorities for care delivery.

The research team will test alternative designs of performance feedback that vary on the following dimension:

1) targets for comparison of one's own performance

The research team will provide feedback on performance by measures that the organization already tracks internally and uses for performance improvement. These include a provider's utilization of opportunities to provide flu vaccinations.

The study will randomly assign different designs of feedback to providers. In order to understand which designs of feedback have the best effects on performance, the research team will test the following hypotheses:

1. Displaying the next-highest quartile will motivate improvement more than display of all quartiles.

   Theory: The next-highest quartile will serve as an injunctive norm, or suggested target, to repeatedly lift an individual's performance to the suggested level.
2. The positive effect of displaying the next-highest quartile, relative to displaying all quartiles, will be most pronounced for initially low performers.

   Theory: The next highest quartile averts upward social comparison to a much higher level of peer performance, which can be discouraging and so negatively affect performance
3. The positive effect of displaying the next-highest quartile, relative to displaying all quartiles, will diminish over time.

   Theory: Individuals may become worn out as they see a target ratchet higher when their performance improves.
4. Displaying team relative performance along with individual relative performance will be more effective than displaying either type of information alone.

ELIGIBILITY:
Inclusion Criteria:

A healthcare provider practicing at The Southeast Permanente Medical Group in a specialty for which the performance measure being studied is relevant.

Health care providers include:

Physicians, Nurse Practitioner, Certified Nurse Midwife, Psych Nurse Specialist, Optometrist, Podiatrist, and Physician Assistant

Exclusion Criteria:

Non-Physicians: Registered Nurses excluding nurse practitioners

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Flu Vaccination Administered During Encounter | 10 Weeks
  Whether or not the providers succeeded in administering flu vaccination during flu vaccination opportunity

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Georgia Regional Offices, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04579614/Prot_SAP_000.pdf